CLINICAL TRIAL: NCT00125372
Title: A Clinical and Pharmacologic Study of the Combination of Erlotinib and Bexarotene in Resectable Clinical Stage I-II Non-Small Cell Lung Cancer
Brief Title: Study of Tarceva and Targretin in Stage I-II Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Ligand Pharmaceuticals (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Konstantin Dragnev, Associate Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-0453
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Carcinoma, Non-small-cell Lung
Keywords: tarceva; targretin; non-small cell lung cancer; carcinoma, non-small cell lung cancer; nsclc
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — Erlotinib Hydrochloride; Bexarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib and Bexarotene (Experimental): Erlotinib 150 mg and bexarotene 400 mg/m2/day will be administered orally for 7 to 9 days prior to thoracotomy.
  Interventions: Drug: erlotinib (Tarceva) and bexarotene (Targretin)

INTERVENTIONS:
Drug: erlotinib (Tarceva) and bexarotene (Targretin) — Erlotinib 150 mg and bexarotene 400 mg/m2/day will be administered orally for 7 to 9 days prior to thoracotomy
  Other Names: Tarceva; Targretin

SUMMARY:
The purpose of this study is to learn the effects on lung cancer of 2 new drugs, Tarceva and Targretin, given in combination before surgical removal of the tumor. Tarceva is approved by the Food and Drug Administration (FDA) for lung cancer. Targretin is approved for the treatment of cutaneous T-cell lymphoma. This combination of drugs is experimental.

DETAILED DESCRIPTION:
Erlotinib 150mg and bexarotene 400mg/m2 will be administered orally for 7-9 days prior to thoracotomy. Plasma samples will be collected on the day before surgery and along with tissue samples on the day of the thoracotomy. Analyses will be done on the resected specimen and it will be compared to the pre-study diagnostic specimen.

ELIGIBILITY:
Inclusion Criteria:

* Resectable stage I or II non-small-cell lung cancer
* Prior tissue biopsy (not cytology) available for research analysis
* Adequate hepatic and renal function

Exclusion Criteria:

* Prior chemotherapy or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin H Dragnev, MD, Principal Investigator — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib and Bexarotene
Started | 12
Completed | 10
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib and Bexarotene
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10
Smoking status [Count of Participants; unit: Participants]
  Current | 3
  Never | 1
  Former | 6
Histology [Count of Participants; unit: Participants]
  Sqamous Cell carcinoma | 1
  Adenocarcinoma | 6
  Adenosquamous carcinoma | 1
  Bronchioloalveolar carcinoma | 1
  Basaloid carcinoma | 1
EGFR Status [Count of Participants; unit: Participants]
  Wild Type | 8
  Mutant | 1
  Not assessed | 1
KRAS Status [Count of Participants; unit: Participants]
  Wild type | 4
  Mutant | 5
  Not assessed | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Change in Expression Level of EGFR.
Time Frame: Baseline and 9 days
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib and Bexarotene
Number analyzed (Participants) | 10
Participants
  Reduction in EGFR expression | 3
  No change | 7

2. Primary Outcome: Number of Participants With Change in Expression Level of Cyclin D1
Time Frame: Baseline and 9 days
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib and Bexarotene
Number analyzed (Participants) | 10
Participants
  Reduction in Cyclin D1 expression | 6
  No change | 4

3. Primary Outcome: Number of Participants With Change in Expression Level of Phosphorylated EGFR (pEGFR)
Time Frame: Baseline and 9 days
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib and Bexarotene
Number analyzed (Participants) | 10
Participants
  Reduction in pEGFR expression | 6
  No change | 4

4. Secondary Outcome: Tumor Tissue Concentrations of Erlotinib and Bexarotene and Correlation With Plasma Levels
Time Frame: At 9 days
Population: The testing necessary to determine the correlation documented in this outcome was not performed due to budget constraints.
Arm/Group | Erlotinib and Bexarotene
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With EGFR Mutations and Correlation of EGFR Mutations With Response
Time Frame: Baseline and 9 days
Population: The numbers analyzed are represented in the rows by EGFR status at baseline. Eight participants had wild-type EGFR at baseline, one had a mutation at Exon 21, and one participant's EGFR status was not assessed at baseline. The total of all rows matches the overall number analyzed; 10.
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib and Bexarotene
Number analyzed (Participants) | 10
Participants
  Wild-type EGFR: number analyzed (Participants) | 8
  Wild-type EGFR: Therapeutic Response | 4
  Wild-type EGFR: No Therepeutic Response | 4
  EGFR Mutation at Exon 21: number analyzed (Participants) | 1
  EGFR Mutation at Exon 21: Therapeutic Response | 1
  EGFR Mutation at Exon 21: No Therepeutic Response | 0
  EGFR not assessed at baseline: number analyzed (Participants) | 1
  EGFR not assessed at baseline: Therapeutic Response | 0
  EGFR not assessed at baseline: No Therepeutic Response | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each patient at the start of study treatment until 4 weeks following surgical resection. The total time of adverse event collection over the course of the study from the first treated subject to the last treated patient's end-of-study visit was 4 years.
Arm/Group | Erlotinib and Bexarotene
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No